CLINICAL TRIAL: NCT03966950
Title: Use of Melatonin for Prevention of POCD After TURP Surgery Under Spinal Anesthesia for Elderly Patients
Brief Title: Use of Melatonin for Preventing POCD in Transurethral Prostate Resection Under Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria José Carvalho Carmona, professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: melatonin POCD
Record Dates: First submitted 2019-05-14; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Melatonin; Cognitive Dysfunction; Postoperative Complications; Prostate Hyperplasia
Keywords: Melatonin; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Complications; Prostatic Hyperplasia | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: randomized, parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melatonin group (Experimental): for the melatonin group, 10 mg of melatonin will be taken per os in the evening before the surgery and in the immediate postoperative night and the first and second postoperative days.
  Interventions: Dietary Supplement: melatonin
- placebo group (Placebo Comparator): For the placebo group, placebo will be administered per os in the evening before the surgery and in the immediate postoperative night and the first and second postoperative days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Dietary Supplement: melatonin — melatonin 10 mg per os in the preoperative night and the immediate postoperative night and the first and second postoperative nights.
  Arms: melatonin group
Drug: Placebo oral tablet — placebo taken per os in the preoperative night and the immediate postoperative night and the first and second postoperative nights
  Arms: placebo group

SUMMARY:
This study aims to evaluate the possible effect of melatonin on prevention of cognitive dysfunction in the postoperative period of elderly patients undergoing transurethral resection of the prostate (TURP) under spinal anesthesia

DETAILED DESCRIPTION:
TURP is the most common surgical procedure performed on male patients over 60 years of age to treat benign prostatic hyperplasia.

One of the concerns, since it compromises the quality of life, is postoperative cognitive dysfunction. It can be due to TURP Syndrome or to other causes, like changing the routine and circadian rhythm for patients with more susceptibility.

The investigators postulate that melatonin premedication and use during the perioperative period could avoid cognitive impairment in patients undergoing TURP surgery that didn't develop major complications, like TURP Syndrome.

Since anesthestic technic could also influence the outcome of POCD, only patients undergoing spinal anesthesia were included in the study,

ELIGIBILITY:
Inclusion Criteria:

patients over 60 years who underwent elective surgery for transurethral prostate ressection under spinal anesthesia.

MME > 18 (for those who had less than 4 years of formal education ) or MME > 23 (for those with 4 or more years of formal education)

Exclusion Criteria:

MME < 18 (for those who had less than 4 years of formal eduaction) or 23 (for those with 4 years or more of formal eduacation); History of cancer, brain disease, seizure, Parkinson, dementia, hallucination or any disorder that affects cognition before the surgery.

Lack of proficiency in portuguese mild or severe hearing loss or blindness.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-11-26 (Estimated); Study Completion 2021-11-26 (Estimated)

PRIMARY OUTCOMES:
early postoperative cognitive dysfunction | 30 days
  a full battery of neuropsychological tests including FOME (Fuld Object memory evaluation test), Stroops colours world test, Trail making test and Wais-III were applied in the preoperative day and compared to the 30-postoperative day evaluation. A z score decline higher than 0,5 in two different domains defines an early postoperative cognitive dysfunction

SECONDARY OUTCOMES:
late postoperative cognitive dysfunction | 180 days
  neuropsychological testings (WAIS - III, Trail Making Test, Stroop Colours Word Test and Fuld Object Memory Evaluation Test) were applied after 6 months of the surgery and the z score is compared to the preoperative evaluation- a z score decline higher than 0,5 in two different domains can define a late postoperative cognitive dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Maria JC Carmona, PHD, Principal Investigator — Associate Professor
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kotekar N, Kuruvilla CS, Murthy V. Post-operative cognitive dysfunction in the elderly: A prospective clinical study. Indian J Anaesth. 2014 May;58(3):263-8. doi: 10.4103/0019-5049.135034. PMID 25024467
- [Result] Kotekar N, Shenkar A, Nagaraj R. Postoperative cognitive dysfunction - current preventive strategies. Clin Interv Aging. 2018 Nov 8;13:2267-2273. doi: 10.2147/CIA.S133896. eCollection 2018. PMID 30519008
- [Result] Segal-Gidan F. Postoperative confusion in older adults. JAAPA. 2017 Apr;30(4):12-16. doi: 10.1097/01.JAA.0000513345.29384.39. PMID 28282301
- [Result] Strom C, Rasmussen LS, Sieber FE. Should general anaesthesia be avoided in the elderly? Anaesthesia. 2014 Jan;69 Suppl 1(Suppl 1):35-44. doi: 10.1111/anae.12493. PMID 24303859
- [Result] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Result] Becher KF. [Delirium in geriatric urology patients]. Urologe A. 2019 Apr;58(4):398-402. doi: 10.1007/s00120-019-0887-4. German. PMID 30859233
- [Result] Fan Y, Yuan L, Ji M, Yang J, Gao D. The effect of melatonin on early postoperative cognitive decline in elderly patients undergoing hip arthroplasty: A randomized controlled trial. J Clin Anesth. 2017 Jun;39:77-81. doi: 10.1016/j.jclinane.2017.03.023. Epub 2017 Mar 31. PMID 28494914
- [Result] Cardinali DP, Furio AM, Brusco LI. The use of chronobiotics in the resynchronization of the sleep/wake cycle. Therapeutical application in the early phases of Alzheimer's disease. Recent Pat Endocr Metab Immune Drug Discov. 2011 May;5(2):80-90. doi: 10.2174/187221411799015354. PMID 22074583
- [Result] Spinedi E, Cardinali DP. Neuroendocrine-Metabolic Dysfunction and Sleep Disturbances in Neurodegenerative Disorders: Focus on Alzheimer's Disease and Melatonin. Neuroendocrinology. 2019;108(4):354-364. doi: 10.1159/000494889. Epub 2018 Oct 28. PMID 30368508
- [Result] Marra A, McGrane TJ, Henson CP, Pandharipande PP. Melatonin in Critical Care. Crit Care Clin. 2019 Apr;35(2):329-340. doi: 10.1016/j.ccc.2018.11.008. Epub 2019 Jan 30. PMID 30784613
- [Derived] Madsen BK, Zetner D, Moller AM, Rosenberg J. Melatonin for preoperative and postoperative anxiety in adults. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD009861. doi: 10.1002/14651858.CD009861.pub3. PMID 33319916